CLINICAL TRIAL: NCT00845104
Title: A Phase II Study of Fludarabine (F), Rituxan (R) and Avastin (A) Followed by RA Maintenance in Patients With Relapsed/Refractory B-cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: Fludarabine Phosphate, Rituximab, and Bevacizumab in Treating Patients With B-Cell Chronic Lymphocytic Leukemia That Has Relapsed or Not Responded To Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Responsible Party: Pagel, John, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2278.00; NCI-2010-00316
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Rituximab; Bevacizumab; Flow Cytometry; Polymerase Chain Reaction; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Drug: fludarabine phosphate; Biological: rituximab; Biological: bevacizumab; Other: laboratory biomarker analysis; Other: flow cytometry; Genetic: polymerase chain reaction; Genetic: fluorescence in situ hybridization

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Biological: rituximab — Given IV
  Other Names: C2B8 Monoclonal Antibody; IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine phosphate, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab and bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving fludarabine phosphate together with rituximab and bevacizumab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving fludarabine phosphate together with rituximab and bevacizumab works in treating patients with B-cell chronic lymphocytic leukemia that has relapsed or not responded to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate PFS at 2 years after FR plus Avastin (A) induction followed by Rituximab plus Avastin (RA) maintenance therapy for relapsed/refractory CLL patients.

SECONDARY OBJECTIVES:

I. To evaluate response rates after FR-A induction and RA maintenance therapy. II. To eliminate residual disease (documented by flow cytometry and/or PCR) in patients who have achieved a CR after FR-A.

III. To estimate the rate of conversion of PR to CR after FR-A. IV. To determine the safety and pharmacokinetics of FR-A and RA maintenance.

OUTLINE:

INDUCTION THERAPY: Patients receive fludarabine phosphate IV over 20-30 minutes once daily on days 1-5 and rituximab IV once daily on days 4 or 5. Treatment repeats every 35 days for 6 courses in the absence of disease progression or unacceptable toxicity. Beginning on day 8 of course 1, patients also receive bevacizumab IV over 30 minutes. Treatment repeats every 21 days for 9 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving complete response, partial response, or nodular partial response proceed to maintenance therapy.

MAINTENANCE THERAPY: Beginning 2 months after completion of induction treatment, patients receive rituximab IV every 3 months and bevacizumab IV over 30 minutes every 3 weeks. Treatment continues for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

ELIGIBILITY:
Inclusion

* Relapse or refractory chronic Lymphocytic leukemia as defined by the WHO criteria and exhibit active disease requiring treatment as per the NCI working group in CLL
* Disease measurable defined by a combination of lymphocytosis >= 5,000/mm^3 in peripheral blood and lymphocytosis >= 30% in bone marrow
* Confirmed CD20 expression on malignant CLL cells
* ECOG performance status of 0-2
* Life expectancy of at least 6 months
* Documented negative serologic testing for human immunodeficiency virus (HIV), hepatitis B (unless serologically positive due to prior vaccination), and hepatitis C within the year prior to enrollment
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN)
* Total serum bilirubin < 2.5 x ULN
* Serum creatinine < 1.5 x ULN
* Hemoglobin > 8 g/dL
* Absolute neutrophil count (ANC) > 1,000 cells/mm^3
* Platelet count > 50,000/mm^3
* PT/INR and PTT < 1.5 x ULN
* Within 2 weeks prior to registration, patients must have had a urinalysis negative for protein or a 24-hour urine collection demonstrating < 500 mg protein
* If female and of child-bearing potential, have a negative serum pregnancy test within 14 days of enrollment
* If sexually active male or sexually active female of reproductive capability, has agreed to use a medically accepted form of contraception from time of enrollment to completion of all follow-up study visits
* Signed an institutional review board (IRB)-approved informed consent document for this protocol

Exclusion

* Patients must not require sustained support of hematopoietic cytokines or transfusion of blood products
* Presence of acute infection or other significant systemic illness
* Central nervous system involvement by malignancy, history of CVA, or seizure
* Previously received Bevacizumab
* Received transplant or Alemtuzumab within 3 months of enrollment
* Received an investigational agent, systemic corticosteroids, chemotherapy, immunotherapy, biologic therapy, antibody therapy (e.g., Rituximab) and/or radiation therapy within one month of enrollment
* Radiation to > 25% of bone marrow or any radiation therapy within 4 weeks prior to start of therapy
* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 6 months
* Fludarabine-refractory disease (no response of disease to >= 3 cycles of a fludarabine-based regimen or relapse within 6 months of fludarabine-based regimen)
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Patients with prior malignancy other than lymphoma, except for adequately-treated skin cancer (basal cell or squamous cell carcinoma), in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years unless approved by the PI
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to Day 1
* History of stroke or transient ischemic attack within 6 months prior to Day 1
* Known CNS disease, except for treated brain metastasis; Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1
* History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria as demonstrated by a UPC ratio >= 1.0 at screening
* Known hypersensitivity to any component of bevacizumab
* Pregnancy (positive pregnancy test) or lactation; use of effective means of contraception (men and women) in subjects of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01

PRIMARY OUTCOMES:
Progression-free survival | At 2 years

SECONDARY OUTCOMES:
Response (complete, partial, or nodular partial response, progressive disease, stable disease, or minimal residual disease) | At 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Pagel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium